CLINICAL TRIAL: NCT02646228
Title: Establishment of Patient Derived Cancer Cell Models to Interrogate Novel Molecular Targets in Metastatic Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jeeyun Lee, MD,PhD,Division of hematology-oncology,Department of medicine, Samsung Medical Center
Other Study IDs: 2015-12-154
Record Dates: First submitted 2016-01-03; First posted 2016-01-05 (Estimated); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Metastatic Cancer
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- molecular profiling, patient derived cells
  Interventions: Other: molecular profiling, patient derived cells

INTERVENTIONS:
Other: molecular profiling, patient derived cells — molecular profiling,patient derived cells sample and experimental methods-Blood sample,tumor tissue or primary cultures of human effusions.
  Malignant ascites, pleural effusions, or pericardial effusions will be collected from patients with metastatic cancer.

SUMMARY:
With rapid advances in molecular oncology, the availability of preclinical in vitro cell models and in vivo animal models with specific genomic aberrations is critical for improved prediction of clinical outcomes in cancer patients. One of the most widely used preclinical models is conventional cell lines, such as the NCI-60 panel of cell lines;these cell lines are widely used in preclinical testing for novel targeted drugs, partially owing to the low expense and reduced labor associated with cell culture compared with other preclinical models, such as animal xenografts. However, recent studies have shown that accumulation of genetic aberrations in cancer cell lines occurs with increasing passage number. These models also lack the heterogeneity of tumors and do not exhibit a proper microenvironment, highlighting the limitations of cell-based models. Consistent with this, Johnson et al. demonstrated that in vivo activities of the cell lines within the NCI-60 panel did not closely correlate with corresponding human cancers.

Therefore, to better preserve the genomic integrity and tumor heterogeneity observed in patients, patient-derived xenograft (PDX) models are being used more frequently. PDX is generated by directly transplanting freshly resected patient tumors into immunocompromised murine hosts with or without an intermediate in vitro culture step. This PDX model is an improvement over cell lines because it can provide both an appropriate tumor microenvironment and heterogeneity of tumor cells. However, the engraftment success rates and growth rates of implanted tumors are highly variable depending on the tumor type, possibly due to insufficient numbers of hematopoietic cells and/or ineffective microenvironmental cues in the mouse stroma. The extent to which tumor cells from freshly resected tumors are able to withstand mechanical stresses and xenotransplantation barriers is also unclear. Furthermore, the use of PDX models for application in clinical oncology is limited owing to the time required for PDX establishment (> 4 months) since most patients with refractory cancer live less than 1 year. Recently, PDC line models have been suggested as an alternative preclinical model to be used as a prediction tool for preclinical drug sensitivity.

Therefore, in this study, the investigators aimed to overcome these potential barriers of pre-existing models by examining the capacity of PDC line models to recapitulate the histological and genomic features of primary patient tumors. In selected cases, the investigators screened drug sensitivity in vitro using PDC lines and compared the results with real-life clinical treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years.
* Patients with histologically confirmed cancer
* Written informed consent form
* Presence of metastatic lesion(s) not amenable to surgical treatment and having malignant effusion in the body cavity which needed to be drained by percutaneous methods for therapeutic purpose.

Exclusion Criteria:

* Concurrent disease or condition that would make the subject inappropriate for study participation or any serious medical condition that would interfere with the subject's safety.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: inclusion criteria are as follows: age ≥ 18 years; pathologically confirmed solid cancer; presence of metastatic lesion(s) not amenable to surgical treatment and having malignant effusion in the body cavity which needed to be drained by percutaneous methods for therapeutic purpose.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-02-04 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
molecular screening(collected of blood,tumor tissue Malignant ascites, pleural effusions, or pericardial effusions will be analyzed) | At the time of study entry.
  To determine the feasibility of the use of patient derived tumor cell models - molecular profiling to direct targeted therapies in the treatment of refractory solid tumors
The success rate of patient derived tumor cell model establishment | 2 years

SECONDARY OUTCOMES:
Progression free survival | 2 years
Duration of response | 2 years
Overall survival | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, Korea, South Korea